CLINICAL TRIAL: NCT03679754
Title: Protocol ATI001-102 Expansion Substudy: Evaluation of Ad-RTS-hIL-12 + Veledimex in Subjects With Recurrent or Progressive Glioblastoma
Brief Title: Evaluation of Ad-RTS-hIL-12 + Veledimex in Subjects With Recurrent or Progressive Glioblastoma, a Substudy to ATI001-102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI001-102 EXP Substudy 2.0
Record Dates: First submitted 2018-08-29; First posted 2018-09-20 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — veledimex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ad-RTS-hIL-12 + veledimex (Experimental): Intratumoral Ad-RTS-hIL-12 and oral veledimex
  Interventions: Biological: Ad-RTS-hIL-12; Drug: veledimex

INTERVENTIONS:
Biological: Ad-RTS-hIL-12 — * 2.0 x 10^11 viral particles (vp) per injection
  * intratumoral injection of Ad-RTS-hIL-12
Drug: veledimex — * 20mg/day
  * 15 oral daily doses of veledimex

SUMMARY:
This research study involves an investigational product: Ad-RTS-hIL-12 given with veledimex for production of human IL-12. IL-12 is a protein that can improve the body's natural response to disease by enhancing the ability of the immune system to kill tumor cells and may interfere with blood flow to the tumor.

The main purpose of this study is to evaluate the safety and tolerability of a single intratumoral injection of Ad-RTS-hIL-12 given with oral veledimex.

DETAILED DESCRIPTION:
Patients who are scheduled for craniotomy and tumor resection will receive one dose of veledimex before the resection procedure. Ad-RTS-hIL-12 will be administered by free-hand injection. Patients will continue on oral veledimex for 14 days.

The study is divided into three periods: the screening period, the treatment period and the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥18 and ≤75 years of age
* Provision of written informed consent for tumor resection, tumor biopsy, samples collection, and treatment with investigational products prior to undergoing any study specific procedures
* Histologically confirmed glioblastoma
* Evidence of supratentorial tumor recurrence/progression by magnetic resonance imaging (MRI) according to Response Assessment in Neuro-Oncology (RANO) criteria after standard initial therapy
* Previous standard-of-care antitumor treatment including surgery and/or biopsy and chemoradiation. At the time of registration, subjects must have recovered from the toxic effects of previous treatments as determined by the treating physician. The washout periods from prior therapies are intended as follows: (windows other than what is listed below should be allowed only after consultation with the Medical Monitor)

  1. Nitrosureas: 6 weeks
  2. Other cytotoxic agents: 4 weeks
  3. Antiangiogenic agents: 4 weeks (NOTE: short use (< 4 doses) of bevacizumab for controlling edema is allowed)
  4. Targeted agents, including small molecule tyrosine kinase inhibitors: 2 weeks
  5. Vaccine-based therapy: 3 months
* Able to undergo standard MRI scans with contrast agent before enrollment and after treatment
* Karnofsky Performance Status ≥70
* Adequate bone marrow reserves and liver and kidney function, as assessed by the following laboratory requirements:

  1. Hemoglobin ≥9 g/L
  2. Lymphocytes >500/mm3
  3. Absolute neutrophil count ≥1500/mm3
  4. Platelets ≥100,000/mm3
  5. Serum creatinine ≤1.5 x upper limit of normal (ULN)
  6. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x ULN. For subjects with documented liver metastases, ALT and AST ≤5 x ULN
  7. Total bilirubin <1.5 x ULN
  8. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) within normal institutional limits
* Male and female subjects must agree to use a highly reliable method of birth control (expected failure rate <5% per year) from the Screening Visit through 28 days after the last dose of study drug. Women of childbearing potential (perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential) must have a negative pregnancy test at screening

Exclusion Criteria:

* Previous treatment with bevacizumab for their disease (NOTE: short use (< 4 doses) of bevacizumab for controlling edema is allowed)
* Subjects receiving systemic corticosteroids during the previous 4 weeks
* Radiotherapy treatment within 4 weeks of starting veledimex
* Subjects with clinically significant increased intracranial pressure (eg, impending herniation or requirement for immediate palliative treatment) or uncontrolled seizures
* Known immunosuppressive disease, or autoimmune conditions, and/or chronic viral infections (eg, human immunodeficiency virus [HIV], hepatitis)
* Use of systemic antibacterial, antifungal, or antiviral medications for the treatment of acute clinically significant infection within 2 weeks of first veledimex dose. Concomitant therapy for chronic infections is not allowed. Subjects must be afebrile prior to Ad-RTS-hIL-12 injection; only prophylactic antibiotic use is allowed perioperatively
* Use of enzyme-inducing antiepileptic drugs (EIAED) within 7 days prior to the first dose of study drug. Note: Levetiracetam (Keppra®) is not an EIAED and is allowed
* Other concurrent clinically active malignant disease, requiring treatment, with the exception of non-melanoma cancers of the skin or carcinoma in situ of the cervix or nonmetastatic prostate cancer
* Nursing or pregnant females
* Prior exposure to veledimex
* Use of medications that induce, inhibit, or are substrates of CYP4503A4 within 7 days prior to veledimex dosing without consultation with the Medical Monitor
* Presence of any contraindication for a neurosurgical procedure
* Unstable or clinically significant concurrent medical condition that would, in the opinion of the Investigator or Medical Monitor, jeopardize the safety of a subject and/or their compliance with the protocol. Examples may include, but are not limited to, colitis, pneumonitis, unstable angina, congestive heart failure, myocardial infarction within 2 months of screening, and ongoing maintenance therapy for life-threatening ventricular arrhythmia or uncontrolled asthma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes Holland, Study Director — Alaunos Therapeutics
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - NYU - Langone Health, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Ad-RTS-hIL-12 + Veledimex: Intratumoral Ad-RTS-hIL-12 and oral veledimex
  Ad-RTS-hIL-12:
  - intratumoral injection of Ad-RTS-hIL-12
  veledimex: - 20mg/day
  - 15 oral daily doses of veledimex
Period: Overall Study
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Started | 36
Completed | 35
Not Completed | 1
Not completed — Investigator request | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS): Overall Safety Population (OSP) includes all subjects who have received at least one dose of veledimex (pretumor resection and) and/or all subjects who received Ad-RTS-hIL-12.
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: Years] | 52.1 [20.8 to 72.40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 5
Height [Median (Full Range); unit: cm] | 172.70 [154.90 to 195.60]
Weight [Median (Full Range); unit: kg] | 76.6 [53.1 to 112.9]

OUTCOME MEASURES:

1. Primary Outcome: Safety of Intratumoral Ad-RTS-hIL-12 and Oral Veledimex in Subjects With Recurrent or Progressive Glioblastoma Based on Evaluation of Adverse Events Summarized by Incidence, Intensity and Type of Adverse Event.
Description: Evaluation of adverse events as assessed by CTCAE v4.03. Adverse events will be summarized based on the incidence, intensity and type of adverse event.
Time Frame: From the first dose of study treatment until 30 days after the last dose of veledimex, lasting approximately 5 months.
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
participants
  Any TEAEs | 36
  Any Serious TEAEs | 10
  Any TEAEs with Toxicity Grade ≥ 3 | 16
  Any TEAEs Leading to Treatment Dose Modification | 11
  Any TEAEs Leading to Treatment Discontinuations | 1
  Any TEAEs Leading to Death | 0
  Any Drug-Related TEAEs | 24
  Any Drug-Related Serious TEAEs | 4
  Any Drug-Related TEAEs with Toxicity Grade ≥ 3 | 8
  Any Drug-Related TEAEs Leading to Treatment Dose Modification | 9
  Any Drug-Related TEAEs Leading to Treatment Discontinuations | 1
  Any Drug-Related TEAEs Leading to Death | 0

2. Primary Outcome: Tolerability of Intratumoral Ad-RTS-hIL-12 and Oral Veledimex in Subjects With Recurrent or Progressive Glioblastoma Will be Assessed Based on Expected Dose Compliance
Description: The Day 0 (as applicable), and Day 1 doses of veledimex were administered by study personnel at the study center.
  Thereafter, subjects could self-administer the remaining once daily dose of veledimex. Subjects were instructed to document veledimex dosing compliance in a subject diary, including the time each dose was taken, the time the subject ate the last meal prior to administration of veledimex, the number of capsules taken, whether the subject missed any veledimex doses, and reason for any missed doses. Investigational product container(s) with any remaining capsules were returned to the study staff on Day 15, and staff assessed dose compliance.
Time Frame: Days 1 through 14 of each 21-day treatment cycle, over a total treatment period of up to 6 cycles (approximately 4 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
Participants
  100% Compliance | 22
  Less than 100% Compliance | 14

3. Secondary Outcome: Determine the Overall Survival (OS) of Ad-RTS-hIL-12 + Veledimex
Description: OS is defined as the duration of time from the first dose of study drug (Day 0) to the date of death from any cause in days or months. Subjects are censored based on the last date known to be alive. For example:
  * Subjects who discontinue the study without documentation of additional follow-up will be censored at the date of discontinuation.
  * Subjects who are lost to follow-up will be censored at last follow-up contact date.
  * Subjects still alive up to 2 years from the first dose of study drug are classified as censored and as having completed all follow-up scheduling.
Time Frame: From the first dose of study drug for up to 2 years.
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP is used for analysis of overall survival.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
Months | 10.68 [7.28 to 20.67]

4. Secondary Outcome: Veledimex Pharmacokinetic Profile: Maximum Plasma Concentration (Cmax)
Description: The maximum plasma concentration (Cmax) of veledimex
Time Frame: 15 days
Population: All Subjects with available plasma-time concentration data post dose on Day 14 and predose on Day 15 are included in the PK Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 17
ng/mL | 68.69 (41.95)

5. Secondary Outcome: Veledimex Pharmacokinetic Profile: Time to Maximum Plasma Concentration (Tmax)
Description: Time to maximum plasma concentration (Tmax) of veledimex. Tmax was estimated based on time of maximum concentration (Cmax) from predose (Day 0 or 14) to predose the following day (Day 1 or 15).
Time Frame: 15 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 17
hr | 4.00 (1.16)

6. Secondary Outcome: Veledimex Pharmacokinetic Profile: Half-life (t1/2)
Description: Half-life (t1/2) of veledimex
Time Frame: 15 days
Population: All subjects with available plasma-time concentration data post dose (steady state) on Day 14 and predose on Day 15 are included in the PK Population.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 17
hr | 16.4 (19.4)

7. Secondary Outcome: Veledimex Pharmacokinetic Profile: Area-under-the-concentration Versus Time Curve (AUC)
Description: Area-under-the-concentration versus time curve (AUC) of veledimex from Day 14 predose to Day 15 predose. AUC was estimated using the elimination rate constant k, where k = ln(Cmax/Ctrough)/time difference and AUC is approximately Cmax/k.
Time Frame: 15 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 17
ng*hr/mL | 771.4 (364.5)

8. Secondary Outcome: Veledimex Pharmacokinetic Profile: Volume of Distribution (Vd)
Description: Volume of distribution (Vd) of veledimex. Vd was calculated using AUC approximated as described in the Outcome Measure Description for Outcome Measure 6.
Time Frame: 15 days
Population: The PK blood sample collection was performed either pre-dose or 3-5 hours post-dose, therefore only Cmax and Ctrough will be summarized and plotted. There will be no parameters including time to maximum plasma concentration (Tmax), half-life (t1/2), area under the curve (AUC), volume of distribution (Vd), and clearance (CL).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 17
mL | 683 (613)

9. Secondary Outcome: Veledimex Pharmacokinetic Profile: Clearance (CL)
Description: Clearance (CL) of veledimex. CL was calculated using AUC approximated as described in the Outcome Measure Description for Outcome Measure 6.
Time Frame: 15 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 17
mL/hr | 32.6 (16.2)

10. Secondary Outcome: Veledimex Concentration Ratio Between the Brain Tumor and the Blood
Description: Veledimex concentration ratio was calculated based on the Day 0 tumor and plasma PK results.
Time Frame: Day 0 (at the time of tumor resection)
Population: All Subjects with available serum-time concentration data are included in the PK Population.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
ratio | 0.63 (0.54)

11. Secondary Outcome: Tumor Objective Response Rate (ORR)
Description: For the ORR calculation, responders are defined as those experiencing a confirmed complete response or confirmed partial response. Non-responders are those either with stable or progressive disease. Those subjects that cannot be assessed will be treated as non-responders for the purposes of deriving the percentage of responders and confidence intervals. Overall Response was assessed at multiple timepoints (day 56, week 16, week 24, and week 48) by the study investigators.
  Changes to the original plan for exploration of estimates of efficacy are summarized below.
  • The best overall response (BOR) endpoint was added to the efficacy assessment and reported here.
Time Frame: 48 weeks
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP is to be used for analysis of dose limiting toxicities, overall survival and progression free survival and finding the maximum tolerated dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
Participants
  Complete Response | 1
  Partial Response | 1
  Stable Disease | 27
  Progressive Disease | 6
  Not Evaluable | 0
  No Response | 1
  Missing | 0

12. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS (progression free survival) is the time in months from the first treatment (either veledimex or Ad-RTS-hIL-12) to the first assessment on which the overall response is reported as disease progression. Subjects withdrawing from the study will be censored at their last non progressive disease response assessment. If a subject does not have a non-progressive disease response assessment, the subject will be censored on the date of the first treatment as described above.
Time Frame: From the first dose of study drug for up to 2 years.
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
Days | 52.17 (39.1)

13. Secondary Outcome: Rate of Pseudo-progression (PSP)
Description: PSP Progression free survival was originally defined for determination of PSP requiring confirmation of progression based on RANO/iRANO criteria guidelines.
Time Frame: From the first dose of study drug for up to 2 years.
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP is denoted as the PP population in this uncontrolled setting.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
Participants | 0

14. Secondary Outcome: Changes From Baseline in Cellular Responses Elicited by Ad-RTS-hIL-12 and Veledimex
Description: Evaluation in changes in immune cell population markers, such as CD3 and CD8 in tumor
Time Frame: Baseline and Week 6.
Population: Due to the study's early termination and limited enrollment, a decision was made not to perform the planned immunohistochemistry (IHC) analyses on collected tumor biopsies. Therefore, no data are available for this endpoint, and zero subjects were analyzed. These analyses will not be performed in the future, and data for this outcome measure will not be reported.
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: Ad-RTS-hIL-12 + Veledimex; Test type: Other; Subjects in the Expansion trial did not have biopsies analyzed for cellular responses

15. Secondary Outcome: Peak Serum Concentration of Interleukin-12 (IL-12)
Description: Serum concentrations of IL-12 were measured at multiple timepoints post-dose. For each participant, the peak (maximum) concentration observed from Day 3 through the 30-day follow-up visit was identified. This measure summarizes the mean of those individual peak concentrations.
Time Frame: Samples were collected at Baseline (Day 1), Day 3, Day 8, and Day 15 of Cycle 1, and at the 30-day follow-up visit.
Population: The Evaluable Safety Population (ESP) includes subjects who have received Ad-RTS-hIL-12 and at least one dose of veledimex after Ad-RTS-hIL-12 administration. The ESP is denoted as the Per Protocol population in this uncontrolled setting.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
pg/mL | 20.3 (5.4)

16. Secondary Outcome: Peak Serum Concentration of Interferon-gamma (IFN-γ)
Description: Serum concentrations of IFN-γ were measured at multiple timepoints post-dose. For each participant, the peak (maximum) concentration observed from Day 3 through the 30-day follow-up visit was identified. This measure summarizes the mean of those individual peak concentrations.
Time Frame: Samples were collected at Baseline (Day 1), Day 3, Day 8, and Day 15 of Cycle 1, and at the 30-day follow-up visit
Population: as for outcome 15
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex
Number analyzed (Participants) | 36
pg/mL | 39.3 (27.3)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from the first dose of study treatment for up to 2 years. All other adverse events were collected from the first dose of study treatment until 30 days after the last dose of veledimex (approximately 5 months).
Description: Evaluation will be based on the incidence, intensity, and type of Adverse Events (AEs), Clinically significant changes in the subjects' physical examinations, vital signs, and ECG evaluations, and clinical manifestations relevant to abnormal laboratory values will be captured as AEs.
Arm/Group | Ad-RTS-hIL-12 + Veledimex
All-Cause Mortality (participants affected / at risk) | 4/36
Serious Adverse Events (participants affected / at risk) | 10/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad-RTS-hIL-12 + Veledimex (N=36)
Seizure (Nervous system disorders) | 2 (2)
Aphasia (Nervous system disorders) | 2 (2)
Brain Oedema (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad-RTS-hIL-12 + Veledimex (N=36)
Headache (Nervous system disorders) | 20 (27)
Seizure (Nervous system disorders) | 7 (10)
Aphasia (Nervous system disorders) | 5 (7)
Hemiparesis (Nervous system disorders) | 6 (7)
Encephalopathy (Nervous system disorders) | 3 (4)
Brain oedema (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Cognitive Disorder (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 2 (2)
Speech Disorder (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (2)
Facial Paralysis (Nervous system disorders) | 1 (2)
Cerebrospinal Fluid Retention (Nervous system disorders) | 1 (1)
Facial Paresis (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Pyramidal Tract Syndrome (Nervous system disorders) | 1 (1)
Subdural Hygroma (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (19)
Constipation (Gastrointestinal disorders) | 7 (9)
Vomiting (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 19 (38)
Platelet Count Decreased (Investigations) | 11 (14)
White Blood Cell Count Decreased (Investigations) | 6 (16)
Aspartate Aminotransferase Increased (Investigations) | 6 (9)
Alanine Aminotransferase Increased (Investigations) | 4 (6)
Neutrophil Count Decreased (Investigations) | 4 (8)
Blood Lactate Dehydrogenase Increased (Investigations) | 2 (2)
Amylase Increased (Investigations) | 1 (2)
C-Reactive Protein Increased (Investigations) | 1 (1)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 (1)
Blood Albumin Decreased (Investigations) | 2 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1)
International Normalised Ratio Increased (Investigations) | 2 (2)
Blood Calcium Decreased (Investigations) | 1 (8)
Blood Potassium Decreased (Investigations) | 1 (2)
Blood Bilirubin Increased (Investigations) | 1 (1)
Heart Rate Increased (Investigations) | 1 (1)
Vitamin D Decreased (Investigations) | 1 (1)
White Blood Cell Count Increased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Pyrexia (General disorders) | 8 (13)
Fatigue (General disorders) | 3 (3)
Gait Disturbance (General disorders) | 2 (2)
Pain (General disorders) | 4 (4)
Influenza Like Illness (General disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 10 (12)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Oral Candidiasis (Infections and infestations) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1)
Confusional State (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Abulia (Psychiatric disorders) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (10)
Hypotension (Vascular disorders) | 1 (1)
Hot Flush (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital Oedema (Eye disorders) | 1 (1)
Vision Blurred (Eye disorders) | 2 (2)
Blepharitis (Eye disorders) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1)
Retinal Exudates (Eye disorders) | 1 (1)
Retinal Tear (Eye disorders) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Spinal Muscular Atrophy (Congenital, familial and genetic disorders) | 1 (2)
Hepatic Lesion (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure shall not occur until (i) twenty-four (24) months have elapsed since Sponsor has notified Institution of the completion of the multi-center Study in order for Sponsor to comply with its obligations under 21 CFR 312.53(c)(4), or (ii) after the publication of the multi-center Study data, if the Study is a multi-center Study or Sponsor confirms in writing there will be no multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT03679754/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03679754/SAP_001.pdf